CLINICAL TRIAL: NCT05864443
Title: Surgeons' Mental Distress and Risks After Severe Complications Following Emergency Surgery in China: a Nationwide Cross-Sectional Questionnaire
Brief Title: Surgeons' Mental Distress and Risks After Severe Complications Following Emergency Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Zhongshan-HHY-02
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-05

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Severe complications following emergency surgery — The respondents are limited to surgeons who had previously experienced severe complications following emergency surgery as chief surgeons.

SUMMARY:
Surgeons experience higher levels of work stress, even under normal circumstances. Many can suffer from substantial levels of mental health issues, especially when faced with severe complications. However, due to a variety of reasons, many surgeons are reluctant to disclose mental health issues or seek psychological help.

Patients in need of emergency surgery are usually characterized by critical conditions and high surgical risks. Emergency surgeons always do not have enough time to clearly explain the ins and outs of the disease to the family members of the patients, only tell the key issues and risks that need to be paid attention to during the operation. The tone of the explanation maybe direct and blunt, which also could cause the incomprehension and dissatisfaction of the patients and their families. Due to the lack of communication, although the patient is in critical condition, the family members always think that the disease should be cured after arriving at the hospital. Therefore, once severe complications occur after the operation, the family members often find it difficult to accept the reality. This is also one of the important reasons for medical disputes in emergency surgery.

In addition to delaying patients' recovery courses, severe complications also place enormous pressure on chief surgeons who performed the operations. Such pressures may bring great risks of psychological distress. Surgeons are also the victims when they encounter severe complications following emergency surgery. Their mental distress should not be minimized. Until now, little has been known about the effects of surgical complications on surgeons. In the current study, based on a large-scale questionnaire survey in China, the investigators aimed to investigate incidences of surgeons' mental distress following severe complications after emergency surgery. The investigators also aimed to identify independent risk factors which could help develop strategies to improve the mental well-being of these surgeons after such incidences.

ELIGIBILITY:
Inclusion Criteria:

* Emergency surgeons who experienced severe complications after Emergency Surgery.

Exclusion Criteria:

* Other conditions that do not meet the inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population are limited to surgeons who had previously experienced severe complications following radical gastrectomy as chief surgeons.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Surgeons' mental health | July 01, 2023 to June 30, 2026
  The clinical features collected in the questionnaire relating to the surgeons' mental distress included: i) feeling burnout, anxiety, or depression; ii) avoiding radical gastrectomy or feeling stress, slowing down the process during radical gastrectomy operations; iii) having physical reactions, including heart pounding, trouble breathing, or sweating while recalling; iv) having urges to quit being a surgeon; v) taking psychiatric medications; and vi) seeking psychological counseling. Meeting any one of the above six clinical features was regarded as having mental distress; Meeting ore or two was defined as mild mental distress, and meeting three or more was defined as severe mental distress.

IPD SHARING:
Plan to Share IPD: Undecided